CLINICAL TRIAL: NCT02835872
Title: A Randomized, Double-Blind, Parallel Study to Evaluate the Effects of a Dietary Fiber Ingredient on Blood Lipids in Men and Women
Brief Title: A Study to Evaluate the Effects of Dietary Fiber on Blood Lipids in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tate & Lyle (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO1604
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolemia
Keywords: fiber; cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cellulose control (Placebo Comparator): 3 g Insoluble Fiber (Cellulose)/d contained within drinks and crackers
  Interventions: Other: dietary fiber
- Soluble fiber treatment (Active Comparator): 3 g soluble dietary fiber test ingredient contained within drinks and crackers
  Interventions: Other: dietary fiber

INTERVENTIONS:
Other: dietary fiber — Fiber containing drink mixes and crackers to be consumed with meals (1g fiber/serving) three times per day for a total of 3 g fiber.

SUMMARY:
There is a need to assess the LDL-C-lowering abilities of a dietary fiber ingredient, in order to confirm the product's efficacy. Thus, the objective of this study is to assess the effect of 3g dietary fiber on lowering serum LDL-C in otherwise healthy men and women.

DETAILED DESCRIPTION:
This study will assess the effect of 3g/d dietary fiber ingredient on lowering serum LDL-C in otherwise healthy men and women. Subjects will be generally healthy men and women (approximately equal number of men and women) 21-79 years of age, inclusive, each with a fasting LDL-C level ≥130 mg/dL and <190 mg/dL.

This randomized, controlled, 28-day parallel study will include one screening Visit (Visit 1, Day -14), two baseline visits (Visits 2 and 3; Days -3 and 0) and three test visits (Visits 4, 5, and 6; Days 14, 25, and 28), and two contact reminders (Days 7 and 21).

Study ingredients will be provided in three servings of study products each day. During the study, subjects will be instructed to consume one serving of study product at each mealtime.

The primary outcome variable will be the percent change in LDL-C concentration from baseline (average of Days -3 and 0) to the end of each intervention condition (average of Days 25 and 28).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a generally healthy male or female, 21-79 years of age, inclusive.
2. Subject has a BMI of ≥18.50 and ≤35.00 kg/m2 at Visit 1 (Day -14).
3. Subject has a fasting LDL-C level ≥130 mg/dL and <190 mg/dL at Visit 1 (Day -14) while receiving no drug therapy. One venous retest allowed for screening subjects within ±3% of the target range (i.e., minimum of 126; maximum of 196 mg/dL). In the event that a redraw is necessary, the average of the two LDL-C values (the redraw value and the Visit 1 value) will be used to determine eligibility.
4. Subject has a fasting TG <400 mg/dL at Visit 1 (Day -14). One venous retest allowed for ≥400 mg/dL values.
5. Subject is willing to maintain a stable body weight, follow the dietary recommendations, and maintain usual physical activity throughout the study period.
6. Subject is willing to maintain usual physical activity level throughout the trial.
7. Subject is a non-user of all tobacco and smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, and e-cigarettes) and has no plans to change status during the study period.
8. Subject is a premenopausal female with a history of regular menstrual cycles that range in length from 21 to 35 d, or subject is a post-menopausal female (i.e., has not had regular menstrual cycles for at least one year).
9. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
10. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Subject has diagnosed diabetes mellitus (Type 1 or Type 2) or fasting glucose ≥126 mg/dL at the screening Visit (Visit 1, Day -14).
2. Subject has a history or presence of uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac, hepatic, renal, gastrointestinal, endocrine, hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's patients), psychiatric (including depression and/or anxiety disorders) or biliary disorders.
3. Subject has abnormal laboratory test results of clinical significance at Visit 1 (Day -14), at the discretion of the Clinical Investigator.
4. Subject has a known allergy or sensitivity to any of the ingredients in the study products.
5. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Clinical Investigator.
6. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -14). One re-test will be allowed on a separate day prior to Visit 3 (Day 0), for subjects with abnormal blood pressure.
7. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
8. Subject has had a weight loss or gain >4.5 kg in the 3 months prior to Visit 1 (Day -14).
9. Subject has used any medications which can alter the lipid profile, including but not limited to: statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, niacin (drug form), thyroid hormones, or omega-3 ethyl ester drugs within 4 weeks of Visit 1 (Day -14; Appendix 2).
10. Subject has used any foods or dietary supplement that might alter lipid metabolism, including but not limited to: omega-3 fatty acid supplements (e.g., flaxseed, fish, or algal oils) or fortified foods, sterol/stanol products; dietary fiber supplements (including Metamucil or viscous fiber-containing supplement); red rice yeast supplements; garlic supplements; soy isoflavone supplements; niacin or its analogues at doses >400 mg/d (or others at the discretion of the Clinical Investigator) within 2 weeks of Visit 1 (Day -14; Appendix 2).
11. Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) or programs within 4 weeks prior to Visit 1 (Day -14, Appendix 2).
12. Subject has an active infection or is using antibiotics within 7 d of the baseline visits (Visits 2 and 3; Days -3).
13. Subject is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
14. Subject has a history or presence of diagnosed severe premenstrual syndrome and/or premenstrual dysphoric disorder which could interfere with subject compliance.
15. Subject has initiated or changed use of hormonal contraceptives within 90 d of Visit 1 (Day -14).
16. Subject has been exposed to any non-registered drug product within 30 d prior to visit 1 (Day -14).
17. Subject has participated in a clinical trial within 4 weeks of Visit 1 (Day -14).
18. Subject has a recent history of (within 12 months of screening; Visit 1, Day -14) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
19. Subject has a lifestyle deemed incompatible with the study according to the Clinical Investigator including high level physical activity (defined as more than 6 hours of vigorous physical activity per week)
20. Individual has a condition the Clinical Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in LDL Cholesterol | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change in Total cholesterol | Baseline and 4 weeks
Change in HDL- Cholesterol | Baseline and 4 weeks
Change in Non-HDL- Cholesterol | Baseline and 4 weeks
Change in Triglycerides | Baseline and 4 weeks
Total / HDL Cholesterol Ratio | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share data at this time.